CLINICAL TRIAL: NCT04147039
Title: A Mobile Phone App to Promote Healthy Diet and Physical Activity in 2.5-year-olds - a Randomised Controlled Trial in Primary Child Health Care.
Brief Title: A Mobile Phone App to Promote Healthy Diet and Physical Activity in 2.5-year-olds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Forte (Industry)
Responsible Party: Principal Investigator, Marie Löf, docent, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-02747
Record Dates: First submitted 2019-10-21; First posted 2019-10-31 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receives the MINISTOP 2.0 mobile phone app for 6 months
  Interventions: Behavioral: MINISTOP 2.0
- Control (No Intervention): Receives standard care through primary child health care

INTERVENTIONS:
Behavioral: MINISTOP 2.0 — The MINISTOP 2.0 is a behavioural change program aiming to promote healthier diet and physical activity among 2.5-year-old children. The program consists of features such as information, monitoring and feedback (dietary key variables, physical activity, screen time) and it is built around 13 themes during the 6-month period.
  Arms: Intervention

SUMMARY:
Childhood obesity is still a major global health issue. The preschool age (2-5 years) has been identified as a critical period to intervene, Mobile technology (mHealth) has been successful for weight loss and behavior changes in adults. This proposed randomized controlled trial aims to assess the effectiveness of an 6-month intervention program, the Mobile-based intervention to stop obesity in preschoolers (MINISTOP) 2.0 mobile phone app integrated in primary child health care for parents of children aged 2.5 years. The MINISTOP 2.0 app is built on the previous MINISTOP 1.0 app. Five hundred children will be recruited at their routine visit at 2.5 years of age and after baseline measures randomized to the intervention or control group. In addition, the investigators will assess acceptability, feasibility and appropriateness of the app by parents and primary child health care nurses.

ELIGIBILITY:
Inclusion criteria:

-Children at the routine visit at 2.5-3 years of age at selected primary child health centers in Sweden

Exclusion criteria:

* Children diagnosed with neurological or endocrine diseases
* Children who have a parent suffering from a serious physical or psychological disease making the study too demanding for the family
* Children from families who will not be able to understand the content of the app (i.e. do not speak Swedish, English, Somali or Arabic)

Ages: 24 Months to 38 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 552 (Actual)
Dates: Start 2019-11-02 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Intake of dietary key indicators as assessed by a questionnaire | At the end of the intervention which is six months after baseline
  Intake of dietary indicators such as fruits and vegetables, sweet and savory treats, sugar-sweetened drinks (in portions or grams per day)
Physical activity as assessed by a questionnaire | At the end of the intervention which is six months after baseline
  Time spent on moderate-to-vigorous physical activity, screen time (min/day)

SECONDARY OUTCOMES:
Body mass index | At the end of the intervention which is six months after baseline
  Body weight divided by squared height
Satisfaction and usage of the app as assessed by a questionnaire and interviews | At the end of the intervention which is six months after baseline
  Percentage of users (parents and primary health care nurses) that were satisfied with app, used features in the app
Usage of the app as assessed using the objectively measured activity in the app | At the end of the intervention which is six months after baseline
  Number of recordings and messages read in the app (per time unit such as per week)
Parental self-efficacy to promote healthy diet and physical activity behaviors in their child as assessed by a questionnaire | At the end of the intervention which is six months after baseline
  Derived scores from selected questions from a questionnaire (Parental Self-Efficacy for Promoting Healthy Physical Activity and Dietary Behaviors in Children Scale (PSEPAD) Questionnaire). The minimum value is 0 and the maximum value 10.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Department of Biosciences and Nutrition, Karolinska Institute, Huddinge
  - Linköping University, Linköping

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alexandrou C, Henriksson H, Henstrom M, Henriksson P, Delisle Nystrom C, Bendtsen M, Lof M. Effectiveness of a Smartphone App (MINISTOP 2.0) integrated in primary child health care to promote healthy diet and physical activity behaviors and prevent obesity in preschool-aged children: randomized controlled trial. Int J Behav Nutr Phys Act. 2023 Feb 21;20(1):22. doi: 10.1186/s12966-023-01405-5. PMID 36810069
- [Derived] Henriksson H, Alexandrou C, Henriksson P, Henstrom M, Bendtsen M, Thomas K, Mussener U, Nilsen P, Lof M. MINISTOP 2.0: a smartphone app integrated in primary child health care to promote healthy diet and physical activity behaviours and prevent obesity in preschool-aged children: protocol for a hybrid design effectiveness-implementation study. BMC Public Health. 2020 Nov 23;20(1):1756. doi: 10.1186/s12889-020-09808-w. PMID 33228572